CLINICAL TRIAL: NCT01758224
Title: Cleveland Clinic Research Program: Expiratory Muscle Conditioning Using Functional Magnetic Stimulation for Patients With Multiple Sclerosis
Brief Title: Expiratory Muscle Conditioning in Multiple Sclerosis Using Magnetic Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: W81XWH-11-1-0707
Record Dates: First submitted 2012-12-19; First posted 2013-01-01 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Functional Magnetic Stimulation; Pulmonary Function
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Functional Magnetic Stimulation (Experimental): This group will receive magnetic stimulation of the respiratory (breathing) muscles that may improve the breathing function in subjects with MS. The magnetic stimulation protocol (plan of study) consists of a daily expiratory (breathing out) muscle conditioning program (20 minutes).
  Interventions: Other: Functional Magnetic Stimulation
- Resistive Expiratory Muscle Training (Active Comparator): Participants in this group will perform breathing exercises using a resistive breathing device. The training will take place in the FMS lab. After training, participants will perform the exercise for 20 minutes daily (5days each week for 6 weeks) in their home.
  Interventions: Other: Resistive Expiratory Muscle Training

INTERVENTIONS:
Other: Functional Magnetic Stimulation — The magnetic stimulation protocol (plan of study) consists of a daily expiratory (breathing out) muscle conditioning program (20 minutes). A magnetic coil will be placed on participant's back to stimulate the nerves related to the breathing function. Each stimulation will last two seconds and the time between each stimulation is about half a minute. The training session will begin with low intensity FMS for 20 minutes daily. The FMS stimulation intensity will gradually increase during the 6-week training period.
  Other Names: FMS
  Arms: Functional Magnetic Stimulation
Other: Resistive Expiratory Muscle Training — The REMT training will take place in the FMS lab using a standard resistive breathing device. After training, participants will perform the exercise for 20 minutes daily (5days each week for 6 weeks) in their home. Participants will wear a nose clip when performing the breathing exercise. The exercise protocol will begin with a low resistance level for 20 minutes a day. The resistance level will gradually increase during the 6-week training period.
  Other Names: REMT
  Arms: Resistive Expiratory Muscle Training

SUMMARY:
Multiple sclerosis (MS) is a primary disorder of the central nervous system that may affect motor pathways and cause muscle weakness. Respiratory complications due to respiratory muscle weakness are common in the terminal stages of MS and contribute to mortality in these patients. Respiratory muscle weakness may also impair the performance of coughing and aspiration, pneumonia, or even acute ventilatory failure may ensue. Functional magnetic stimulation (FMS) is a non-invasive method that promotes the contraction of muscles through nerve activation. Over the last few years, the study investigators have demonstrated efficacy of FMS technology for stimulating respiratory muscles in animal models, able-bodied subjects [3] and spinal cord injured (SCI) patients [4]. In this study, the researchers will investigate the efficacy of using FMS technique for respiratory muscle conditioning in patients with MS. Furthermore, the investigators will also compare expiration related outcomes of FMS technique with resistive expiratory muscle training (REMT) methodology.

Hypotheses

1. FMS conditioning of the expiratory muscles can generate significant expiratory flows and pressures in patients with MS.
2. FMS conditioning of expiratory muscles is more effective compared to resistive expiratory muscle training (REMT) in patients with MS.

DETAILED DESCRIPTION:
Optimal respiratory function depends on intact neural circuitry which orchestrates the interplay between respiratory muscles and intrinsic pulmonary function to maintain adequate ventilation. In the absence of respiratory muscle activation, pressure gradients cannot be developed and air exchange at the alveolar surface cannot occur. Thus, any impairment in respiratory muscle performance can lead to pulmonary dysfunction, respiratory distress and even death. Multiple sclerosis (MS) is a primary disorder of the central nervous system that often affects motor pathways, causing diminished muscle strength and endurance throughout the body including the ventilatory muscles. Respiratory complications are recognized as the major cause of morbidity and mortality in individuals with advanced MS. The investigators' research team has over 15 years of experience using Functional Magnetic Stimulation (FMS) for stimulating nerves and muscles below the level of injury in patients with chronic SCI; and has also demonstrated significant benefit for improving respiratory muscles, bladder and bowel functions. In this study, the investigators will investigate the efficacy of using FMS technique for respiratory muscle conditioning in patients with multiple sclerosis; and will compare the results of the expired functions (volume, pressure, and flow) generated by using the FMS technique with data obtained from using the resistive expiratory muscle training (REMT) methodology.

ELIGIBILITY:
Inclusion Criteria:

* Multiple Sclerosis diagnosis
* Baseline maximal expiratory pressure (MEP) values between 50% and 70% of predicted values
* Patients must also be in stable condition and free of active brain disease or cardiovascular disorders (history of myocardial infarction, congestive heart disease, or uncontrolled hypertension).

Exclusion Criteria:

* Cardiac pacemakers, ferromagnetic metal implants, uncontrolled high blood pressure, active pulmonary conditions such as chronic obstructive pulmonary disease, bronchiectasis, asthma, and diaphragmatic paralysis.
* Patients who are ventilator dependent, with significant scoliosis, other chest wall deformity, obesity, severe diabetes mellitus, as well as pregnant women will be excluded from participating in the study.
* Patients with substance abuse or mental incompetence will also be excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Pulmonary Function Testing (PFT) | At study initiation and every two weeks over a 14 week period (8 PFTs)
  Changes in participant's pulmonary (lung) function will be assessed using a non-invasive pulmonary function test (PFT).

CONTACTS AND LOCATIONS:
Overall Officials: Vernon W Lin, MD PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lin VW, Hsiao IN, Zhu E, Perkash I. Functional magnetic stimulation for conditioning of expiratory muscles in patients with spinal cord injury. Arch Phys Med Rehabil. 2001 Feb;82(2):162-6. doi: 10.1053/apmr.2001.18230. PMID 11239305
- [Background] Singh H, Magruder M, Bushnik T, Lin VW. Expiratory muscle activation by functional magnetic stimulation of thoracic and lumbar spinal nerves. Crit Care Med. 1999 Oct;27(10):2201-5. doi: 10.1097/00003246-199910000-00022. PMID 10548207